CLINICAL TRIAL: NCT04022460
Title: Using Personal Mobile Technology to Identify Obstructive Sleep Apnea in Children With Down Syndrome (UPLOAD)
Acronym: UPLOAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Sherri Katz, Chief, Division of Pediatric Respirology, Children's Hospital of Eastern Ontario
Other Study IDs: 19/30X
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea; Child
Keywords: Polysomnography; Pediatric; Down syndrome; Obstructive sleep apnea; Screening tool; Mobile technology
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Video clip assessment — Parents will take short video clips of their child sleeping at night. They will be asked to review the video clips and rate whether they think their child has obstructive sleep apnea (OSA), and if so, how severe it is. Two clinicians will review the video clips on a separate night.
Diagnostic Test: Polysomnography (sleep study) — Children will undergo a polysomnography as the gold standard test to assess for OSA.
Other: Educational webinar — After evaluating the video clips of their child sleeping, parents will watch an educational webinar on OSA in children with Down syndrome and how to recognize symptoms.

SUMMARY:
This study aims to see if mobile video clips (smartphone recordings) can be used to screen children with Down syndrome to identify those at highest risk of obstructive sleep apnea (OSA), so they can be prioritized for an earlier sleep study. Parents will be asked to record short video clips of their child sleeping, and then rate whether they think their child has OSA. Later, children will undergo a sleep study to compare to the ratings.

DETAILED DESCRIPTION:
Children with Down syndrome have approximately a 50% chance of developing obstructive sleep apnea (OSA) in their lifetime. OSA is a serious condition where a person stops breathing periodically during sleep; it is associated with high blood pressure, behavioural issues, and lower quality of life. Early diagnosis and treatment is critical, but the best way to diagnose OSA, a 'sleep study', is in short supply. Given the limited resources, this study aims to see if mobile video clips (smartphone recordings) can be used to screen children with Down syndrome to identify those at highest risk of OSA, so they can be prioritized for an earlier sleep study.

Parents of children with Down syndrome, recruited from clinic, will be asked to record short video clips of their child sleeping. Parents will independently rate whether they think their child has OSA and how severe it is, based on the videos, as will two clinicians. Parents will also watch an educational webinar and be asked to re-rate the presence and severity of OSA in their child, to see if the webinar improves their accuracy. Finally, children will undergo a sleep study to compare to the ratings. This study will help determine whether videos can be used to accurately screen for OSA in this high risk population, prioritizing children for earlier diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome
* Within the catchment area of the Children's Hospital of Eastern Ontario Down Syndrome clinic

Exclusion Criteria:

* Previous diagnosis of sleep-disordered breathing on polysomnography
* No access to mobile technology to record video clips
* Children unable to cooperate for polysomnography
* Caregiver does not speak French or English

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of children with Down syndrome who have not previously been diagnosed with sleep-disordered breathing. We will approach children followed at the CHEO Down Syndrome clinic to participate in this study. All children within CHEO's catchment area will be considered eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Parental screening assessment of presence/absence of OSA based on homemade video clip | 1 day
  Questionnaire developed at CHEO by Pediatric Respirologists and Otolaryngologists. The question of interest is "Do you think your child has obstructive sleep apnea?" The reviewer (a parent) will choose 'Yes' or 'No' after reviewing the homemade video clips. This is a dichotomous outcome with 'Yes' considered as the highest score. The gold standard reference test will be a polysomnography.

SECONDARY OUTCOMES:
Parental assessment of severity of OSA based on homemade video clip | 1 day
  Questionnaire developed at CHEO by Pediatric Respirologists and Otolaryngologists. The question of interest is "Do you believe the severity of the obstructive sleep apnea is: a) Mild, b) Moderate, or c) Severe ?" This question will only appear to parents who chose 'Yes' for the primary outcome. The reviewer will answer the question after reviewing the homemade video clips. This is an ordinal outcome with 'Mild' being considered the lowest score (1), and 'Severe' being considered the highest score (3). The gold standard reference test will be a polysomnography.
Physician screening assessment of presence/absence of OSA based on homemade video clip | 1 day
  Questionnaire developed at CHEO by Pediatric Respirologists and Otolaryngologists. The question of interest is "Do you think your child has obstructive sleep apnea?" Two physicians will independently choose 'Yes' or 'No' after reviewing the homemade video clips. This is a dichotomous outcome with 'Yes' considered as the highest score. The gold standard reference test will be a polysomnography.
Physician assessment of severity of OSA based on homemade video clip | 1 day
  Questionnaire developed at CHEO by Pediatric Respirologists and Otolaryngologists. The question of interest is "Do you believe the severity of the obstructive sleep apnea is: a) Mild, b) Moderate, or c) Severe ?" This question will only appear to physicians who choose 'Yes' for Outcome #3. The reviewer will answer the question after reviewing the homemade video clips. This is an ordinal outcome with 'Mild' being considered the lowest score (1), and 'Severe' being considered the highest score (3). The gold standard reference test will be a polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada